CLINICAL TRIAL: NCT02312908
Title: Effect of Clonazepam on REM Sleep Behavior Disorder in Patients With Parkinsonism: a Prospective, Randomized, Double-blind and Placebo-controlled Trial
Brief Title: Effect of Clonazepam on REM Sleep Behavior Disorder in Patients With Parkinsonism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, BS Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14172EuiYakAn178
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: REM Sleep Behavior Disorder
Keywords: REM Sleep Behavior Disorder; Parkinson Disease; Placebos; Randomized Controlled Trial; Double-Blind Method; Clinical Trial
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease | interventions — Clonazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clonazepam (Experimental): Clonazepam 0.5 mg 1 Tablet by mouth, 1/day before sleeping for 4 weeks
  Interventions: Drug: Clonazepam
- Placebo (Placebo Comparator): Placebo 1 Tablet by mouth, 1/day before sleeping for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonazepam — For experimental treatment of RBD
  Other Names: Rivotril
  Arms: Clonazepam
Drug: Placebo — Placebo pill manufactured to mask clonazepam 0.5mg tablet
  Other Names: Placebo tablet of Rivotril
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether clonazepam is effective and safe in the treatment of rapid eye movement behavior disorder (RBD) of patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
RBD is one of the representative non-motor symptoms of PD and other synucleinopathies. Patients with RBD show dream-enacting behaviors such as punching, kicking, singing, screaming, or somnambulism. These can interfere in sleep quality and increase the risk of falling down from the bed and physical injuries of both the patient and sleep partner. Therefore, qualities of life of the patient and sleep partner are negatively influenced by presence of RBD.

Clonazepam has been used for treatment of choice of RBD. It decreased RBD symptoms completely in 55-79% and partially in 11-32% of patients. However, these results are based on open-label or descriptive studies. There has been no randomized placebo controlled study that evaluated the efficacy and safety of clonazepam for treating RBD.

ELIGIBILITY:
Inclusion Criteria:

* Subject was enrolled voluntarily and understood the contents of this clinical trial
* Subject was diagnosed as Parkinson disease (PD) or Parkinson's syndrome
* Hoehn and Yahr (H&Y) stage 1, 2, or 3
* Existence of caregivers who can provide a information about symptoms of rapid eye movement sleep disorder (RBD) of the participant
* Existence of RBD by answering "yes" to the question (RBD-1Q): "Have you ever been told, or suspected yourself, that you seem to 'act out your dreams' while asleep (for example, punching, flailing your arms in the air, making running movements, etc.)?"

Exclusion Criteria:

* Existence of cognitive decline hard to participate in the clinical trial
* Subject has confusion or visual hallucination in daytime
* Diagnosed as obstructive sleep apnea or severe snoring
* Previous clonazepam treatment within 4 weeks
* Current treatment with benzodiazepines at bedtime
* Alcoholics or drug abuser
* Lactating, pregnant, or possible pregnant
* Hypersensitivity to clonazepam or benzodiazepines
* Prior participation to other clinical trials within 3 months
* Presence of severe comorbidities or a cancer
* Existence of illness or problems which makes difficult to be enrolled to this trial judged by clinicians

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression-Improvement scale (CGI-I) | Four weeks (plus or minus 3 days)
  Clinician assessed rating scale of clinical improvement or worsening relative to a baseline state, scored as 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.

SECONDARY OUTCOMES:
Clinical Global Impression-Severity scale (CGI-S) | Four weeks (plus or minus 3 days)
Epworth Sleepiness Scale (ESS) | Four weeks (plus or minus 3 days)
Parkinson Disease Sleep Scale (PDSS) | Four weeks (plus or minus 3 days)
Montreal Cognitive Assessment (MoCA) | Four weeks (plus or minus 3 days)
Unified Parkinson's Disease Rating Scale (UPDRS) | Four weeks (plus or minus 3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Beom Seok Jeon, MD, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arnulf I. REM sleep behavior disorder: motor manifestations and pathophysiology. Mov Disord. 2012 May;27(6):677-89. doi: 10.1002/mds.24957. Epub 2012 Mar 22. PMID 22447623
- [Background] Sixel-Doring F, Trautmann E, Mollenhauer B, Trenkwalder C. Associated factors for REM sleep behavior disorder in Parkinson disease. Neurology. 2011 Sep 13;77(11):1048-54. doi: 10.1212/WNL.0b013e31822e560e. Epub 2011 Aug 10. PMID 21832215
- [Background] Postuma RB, Bertrand JA, Montplaisir J, Desjardins C, Vendette M, Rios Romenets S, Panisset M, Gagnon JF. Rapid eye movement sleep behavior disorder and risk of dementia in Parkinson's disease: a prospective study. Mov Disord. 2012 May;27(6):720-6. doi: 10.1002/mds.24939. Epub 2012 Feb 9. PMID 22322798
- [Background] Gagnon JF, Postuma RB, Montplaisir J. Update on the pharmacology of REM sleep behavior disorder. Neurology. 2006 Sep 12;67(5):742-7. doi: 10.1212/01.wnl.0000233926.47469.73. PMID 16966533
- [Background] Schenck CH, Hurwitz TD, Mahowald MW. Symposium: Normal and abnormal REM sleep regulation: REM sleep behaviour disorder: an update on a series of 96 patients and a review of the world literature. J Sleep Res. 1993 Dec;2(4):224-231. doi: 10.1111/j.1365-2869.1993.tb00093.x. PMID 10607098
- [Background] Olson EJ, Boeve BF, Silber MH. Rapid eye movement sleep behaviour disorder: demographic, clinical and laboratory findings in 93 cases. Brain. 2000 Feb;123 ( Pt 2):331-9. doi: 10.1093/brain/123.2.331. PMID 10648440
- [Background] Howell MJ, Arneson PA, Schenck CH. A novel therapy for REM sleep behavior disorder (RBD). J Clin Sleep Med. 2011 Dec 15;7(6):639-644A. doi: 10.5664/jcsm.1470. PMID 22171203
- [Background] Aurora RN, Zak RS, Maganti RK, Auerbach SH, Casey KR, Chowdhuri S, Karippot A, Ramar K, Kristo DA, Morgenthaler TI; Standards of Practice Committee; American Academy of Sleep Medicine. Best practice guide for the treatment of REM sleep behavior disorder (RBD). J Clin Sleep Med. 2010 Feb 15;6(1):85-95. PMID 20191945
- [Background] De Cock VC, Vidailhet M, Arnulf I. Sleep disturbances in patients with parkinsonism. Nat Clin Pract Neurol. 2008 May;4(5):254-66. doi: 10.1038/ncpneuro0775. Epub 2008 Apr 8. PMID 18398415
- [Background] Postuma RB, Arnulf I, Hogl B, Iranzo A, Miyamoto T, Dauvilliers Y, Oertel W, Ju YE, Puligheddu M, Jennum P, Pelletier A, Wolfson C, Leu-Semenescu S, Frauscher B, Miyamoto M, Cochen De Cock V, Unger MM, Stiasny-Kolster K, Fantini ML, Montplaisir JY. A single-question screen for rapid eye movement sleep behavior disorder: a multicenter validation study. Mov Disord. 2012 Jun;27(7):913-6. doi: 10.1002/mds.25037. Epub 2012 May 30. PMID 22729987
- [Background] Kunz D, Mahlberg R. A two-part, double-blind, placebo-controlled trial of exogenous melatonin in REM sleep behaviour disorder. J Sleep Res. 2010 Dec;19(4):591-6. doi: 10.1111/j.1365-2869.2010.00848.x. PMID 20561180